CLINICAL TRIAL: NCT05778448
Title: Brain-computer Interface (BCI) Based Closed-loop Training for Hemiparetic Upper Extremities in Patients Due to Stroke: A Randomized Controlled Study
Brief Title: BCI for Hemiparetic Upper Extremities in Patients Due to Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Kenneth N. K. Fong, Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BCI_KennethFong_PabloCruz
Record Dates: First submitted 2023-01-31; First posted 2023-03-21 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Stroke; Brain Computer Interface
Keywords: Stroke; Brain Computer Interface; Neurorehabilitation; Event Related Desynchronization
MeSH Terms: conditions — Stroke | interventions — Brain-Computer Interfaces

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- BCI-FES-VR (Experimental): Participants look at an external screen displaying the VR avatar participant's arms while performing wrist dorsiflexion MI in random order (left or right). The BCI system detects the ERD of the motor area corresponding to correct MI. Then, visual feedback with the VR and motor-tactile feedback with the discharge of the FES is delivered. Each session requires 240 MI trials with a training duration of 10 sessions in a 3-week interval.
  Interventions: Device: Brain Computer Interface/ Functional Electrical Stimulation/ Virtual Reality
- BCI-FES (Active Comparator): Same procedure as arm 1 (BCI-FES-VR), but the difference is that the participant's hands replace the VR system. Each session requires 240 MI trials with a training duration of 10 sessions in a 3-week interval.
  Interventions: Device: Brain Computer Interface/ Functional Electrical Stimulation/ Virtual Reality
- BCI-VR (Active Comparator): Same procedure as arm 1 (BCI-FES-VR), but the FES is removed. Each session requires 240 MI trials with a training duration of 10 sessions in a 3-week interval. Each session requires 240 MI trials with a training duration of 10 sessions in a 3-week interval.
  Interventions: Device: Brain Computer Interface/ Functional Electrical Stimulation/ Virtual Reality

INTERVENTIONS:
Device: Brain Computer Interface/ Functional Electrical Stimulation/ Virtual Reality — A BCI system involves 3 main components - (1) brain activity collection, (2) external devices triggered by specific features of brain activity, and (3) a processor which decodes the brain activity signal and then translates it into computerized commands to control external devices such as virtual games and functional electrical stimulation (FES).

SUMMARY:
Non-invasive brain-computer interface (BCI) technology is one of the new training approaches to achieve motor restoration through a closed-loop system from brain activity through event-related desynchronization (ERD) after motor imagery (MI) or movement attempt to peripheral feedback triggered by an external hepatic device. Often, it is unclear whether the BCI intervention itself or the assistance of the external device leads to neural responses and functional gains.

This study adopts a closed-loop BCI system involving ERD induced by MI. Functional electrical stimulation (FES) and virtual reality (VR) are simultaneously delivered as feedback. The aim is to investigate the efficacy of closed-loop BCI training combined with FES and VR on the recovery of the hemiparetic upper extremity of individuals with chronic stroke.

Chronic stroke survivors are being recruited and randomly allocated into 3 groups: (1) BCI-FES-VR - participants look at an external screen displaying the VR avatar participant's arms while performing wrist dorsiflexion MI in random order (left or right). The BCI system detects the ERD of the motor area corresponding to correct MI. Then, visual feedback with the VR and motor-tactile feedback with the discharge of the FES is delivered; (2) BCI-FES - same procedure as group 1, but the difference is that the participant's hands replace the VR system; (3) BCI-VR - same procedure as group 1, but the FES is removed. Each session requires 240 MI trials with a training duration of 10 sessions in a 3-week interval.

Motor and MI assessments are being conducted at post-assessment and at a 3-week follow-up.

The findings of this study will provide significant new information regarding neurophysiological motor relearning mechanisms, which could inform the development and evaluation of BCI-based treatment for individuals with stroke and impact the field of translational neuroscience.

ELIGIBILITY:
Inclusion Criteria:

1. Have a diagnosis of ischemic or hemorrhagic stroke to unilateral hemisphere, confirmed by neuroimaging examinations, i.e., brain CT or MRI;
2. Chronic phase of stroke, i.e., time after stroke onset more than 6 months;
3. Between 18 and 64 years old;
4. With severe to moderate levels of hemiparetic upper limb impairment due to stroke, i.e., from levels 1 to 4 in the Functional Test for the Hemiplegic Upper Extremity (FTHUE)
5. Able to give informed written consent to participate in the study.

Exclusion Criteria:

1. Previous diagnosis of any neurological disease excluding stroke;
2. Presence of any sign of cognitive problems (Abbreviated Mental Test < 6)
3. Modified Ashworth score > 2 in wrist extensor muscle in the hemiparetic upper extremity after stroke (Bohannon and Smith, 1987) or with severe pain that hinders upper extremity movement
4. With other notable impairments of the upper extremity not caused by stroke (e.g., fracture, Rheumatoid Arthritis, or congenital deformity, etc.)

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-08-11 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Fugl-Meyer Assessment - Upper Extremity (FMA-UE) | Baseline, Post-intervention and 3-week Follow-up (through study completion, an average of 6 weeks)
  FMA-UE is a clinical assessment for upper limb motor impairment after stroke. It includes 33 items assessing the movement, coordination, and reflex actions of the shoulder, elbow, forearm, and wrist, and the hand joints of the hemiparetic arm. Each item consists of a 3-point ordinal scale (0, 1 and 2), with a total score of 66. The higher the score, the better the performance.
Change from Baseline Action Research Arm Test (ARAT) | Baseline, Post-intervention and 3-week Follow-up (through study completion, an average of 6 weeks)
  The ARAT is a clinical assessment for upper limb functional activities for patients with stroke. The ARAT assesses proximal and distal components of upper limb function. It consists of four subscales: grasp, grip, pinch, and gross movement. It has 19 movement tasks, each graded using a four-point ordinal scale (total scores range from 0 to 57)

SECONDARY OUTCOMES:
Revised Purdue Spatial Visualization Test (Revised PSVT:R) | Baseline, Post-intervention and 3-week Follow-up (through study completion, an average of 6 weeks)
  This test consists of 30 questions designed to see how well a participant can visualize the rotation of three-dimensional objects.
  objects. Each correct answer scores 1 point. The total score is 30 points. The higher the score, the better the performance.
Kinesthetic and Visual Imagery Questionnaire (KVIQ) | Baseline, Post-intervention and 3-week Follow-up (through study completion, an average of 6 weeks)
  The aim of this questionnaire is to determine the extent to which individuals are able to visualize and feel imagined movements. All movements are assessed from a sitting position. The questionnaire includes a visual imagery scale and a kinesthetic imagery scale. The long version (KVIQ-20) comprises 20 items (10 movements for each scale). The rating scale is a 5-point ordinal scale, the clarity of the visual image ( Items V1 to V10) or the intensity of the sensations associated with the imagined movement (Items K1 to K10). The higher the score, the better the outcome. The highest score is 50.
Hand grip strength test | Baseline, Post-intervention and 3-week Follow-up (through study completion, an average of 6 weeks)
  It is a measure of muscular strength or the maximum force/tension generated by the participant's forearm muscles.
Motor Activity Log (MAL) | Baseline, Post-intervention and 3-week Follow-up (through study completion, an average of 6 weeks)
  It is a subjective measure of an individual's real life functional upper limb performance and consists of two scales: the amount of use and quality of movement. The MAL adopts a 6-point ordinal scale from 0 to 5. The higher the score, the better the outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- The Hong Polytechnic University, Department of Rehabilitation Sciences, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bai Z, Fong KNK, Zhang JJ, Chan J, Ting KH. Immediate and long-term effects of BCI-based rehabilitation of the upper extremity after stroke: a systematic review and meta-analysis. J Neuroeng Rehabil. 2020 Apr 25;17(1):57. doi: 10.1186/s12984-020-00686-2. PMID 32334608
- [Background] Sitaram R, Ros T, Stoeckel L, Haller S, Scharnowski F, Lewis-Peacock J, Weiskopf N, Blefari ML, Rana M, Oblak E, Birbaumer N, Sulzer J. Closed-loop brain training: the science of neurofeedback. Nat Rev Neurosci. 2017 Feb;18(2):86-100. doi: 10.1038/nrn.2016.164. Epub 2016 Dec 22. PMID 28003656
- [Background] Cruz Gonzalez, P., Fong, K. N., & Brown, T. (2022). Closed-Loop Brain-Computer Interface Training for Hemiparetic Upper Extremities in Patients with Chronic Stroke: A randomized control study [Abstract]. Neurorehabilitation and Neural Repair. Poster presentation at the 12th World Congress for Neurorehabilitation, December 2022, Vienna, Austria.